# **Statistical Analysis Plan**

| Study Title: | Genetic Determinants of the Coronary Microvascular |
|-------------------|----------------------------------------------------|
| | Obstruction in Percutaneous Coronary Interventions |
| Protocol Number: | CMVO-SNP-2022 |
| Study Number: | NCT05355532 |
| Document date and | Version number 1 from April 24, 2022 |
| version: | |
| Sponsor: | Privolzhsky Research Medical University |
| Principal | Principal Investigator: |
| Investigator: | Ilya Grigorievich Pochinka, MD |
| | Research Center: |
| | State Budgetary Healthcare Institution of Nizhny |
| | Novgorod Region "City Clinical Hospital No. 13 of |
| | Avtozavodsky District of Nizhny Novgorod" |
| | Research Center Address: |
| | 51 Patriotov Street, Avtozavodsky District, |
| | Nizhny Novgorod, Russian Federation, 603018 |
| | Research Center Phone: |
| | +7 (831) 255-28-80 |

- 1. Primary Objective: to identify statistically significant associations between selected SNPs and CMVO development post-PCI in STEMI patients.
- 2. Data Preparation
- 2.1 Data Collection
  - Genetic data: SNP genotypes (binary: variant present/absent)
  - Clinical data:
    - demographics
    - o angiographic parameters
    - laboratory values
    - procedural details
    - hospitalization outcomes
    - o CMVO presence/absence

## 2.2Data Cleaning

- Missing data: exclude samples with >10% missing SNP calls.
- Quality control: Hardy-Weinberg equilibrium testing (p<0.05 threshold for exclusion)
- 3. Statistical Methods
- 3.1 Statistical Analysis
  - Univariate analysis:
    - McNemar's test (matched case-control design) for categorical SNPs
    - Odds ratios (OR) with 95% confidence intervals
  - Multivariate analysis:
    - Conditional logistic regression
    - o OR with 95% confidence intervals
- 3.2 Sensitivity Analysis
  - Re-run analysis using dominant/recessive genetic models
- 4. Outcome Measures
  - Primary endpoint: CMVO
  - Secondary endpoints:
    - o In-hospital mortality

- Left Ventricle Ejection Fraction
- Ventricular fibrillation
- o N-terminal Pro-brain Natriuretic Peptide
- o Six-minute Walk Test

### 5. Statistical Software

R

# 6. Sample Size Justification

- 80 patients (40 CMVO+/40 CMVO-) provides:
  - ∘ 80% power to detect OR $\geq$ 4.0 ( $\alpha$ =0.05, two-tailed)
  - Assumes SNP prevalence = 12–69% (average 50%)

### 7. Data Presentation

- Tables:
  - Baseline characteristics (Me [Q1; Q3] for continuous; n (%) for categorical)
  - o SNP frequencies by group
  - Multivariate ORs for CMVO predictors
- Figures:
  - Flowchart of patient inclusion
  - o Forest plot of significant SNPs

## 8. Ethical Considerations

- All analyses will use anonymized data (patient serial numbers only).
- Protocol deviations documented in CONSORT flowchart.
- Approval:

Local Ethics Committee Protocol Version: 1.0